CLINICAL TRIAL: NCT05547737
Title: Multicenter, Prospective, Real World Study of Camrelizumab in Cross-line Treatment of Non-small Cell Lung Cancer
Acronym: NSCLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: NSCLC-RWS-001
Record Dates: First submitted 2022-06-28; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-05

CONDITIONS: NSCLC
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Camrelizumab — Cross - line treatment of Camrelizumab in non-small cell lung cancer

SUMMARY:
To explore the effectiveness and safety of Camrelizumab based cross-line therapy for patients with advanced NSCLC in the real world

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and volunteered to join the study
2. Aged >=18 years
3. Patients with stage IIIb, IV, or relapsed non-small cell lung cancer diagnosed cytologically or histopathologically as EGFR/ALK-
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. At least one measurable lesion (according to RECIST 1.1)
6. No prior systemic therapy for advanced/metastatic NSCLC
7. contraception

Exclusion Criteria:

1. Those who are allergic to drug treatment；
2. Patients who were also treated with other immunodrugs or therapies；
3. Patients who are participating in other intervention studies；
4. Patients with other malignant tumors at the same time；
5. Pregnant or lactating women；
6. The investigator did not consider the patients eligible to participate in the study under any other circumstances.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stage IIIb, IV, or relapsed non-small cell lung cancer diagnosed cytologically or histopathologically as EGFR/ALK-
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-21 (Estimated); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in second-line treatment of patients with non-small cell lung cancer based on Camrelizumab regimen | Up to 12 months
  CR+PR

SECONDARY OUTCOMES:
Evaluation of Progression Free survival (PFS) in patients with non-small cell lung cancer based on first-line/second-line treatment with Camrelizumab | Up to 36 months
  Progression free survival (PFS) according to RECIST 1.1
Evaluation of second progression-free survival (PFS2) in patients with non-small cell lung cancer based on Camrelizumab regimen | Up to 12 months
  Evaluation of second progression-free survival (PFS2) in patients with non-small cell lung cancer based on Camrelizumab regimen
OS | Up to 12 months
  Overall survival
To evaluate the safety of Camrelizumab based first/second line therapy in patients with non-small cell lung cancer | Up to 12 months
  according to NCI-CTCAE version 5.0

IPD SHARING:
Plan to Share IPD: No